CLINICAL TRIAL: NCT03204175
Title: A Randomised Control Trial of a Sanitation Operation and Management Intervention in Elementary Schools in the Philippines (Fit for School Plus)
Brief Title: Fit Plus: Assessing the Impact of a School-based Intervention on Toilet Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Deutsche Gesellshaft fur Internationale Zusammenarbeit (GIZ) GMBH (Unknown); Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12238
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2017-06

CONDITIONS: Hand Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fit Plus (Experimental): The experimental arm will receive the Fit For School expanded intervention, which addresses pupil handwashing, toothbrushing, and school sanitation maintenance. Interventions will begin in July 2017.
  Interventions: Other: FIT Plus
- Comparator (Active Comparator): This group will receive the Fit Plus intervention after the trial is complete (January 2017)
  Interventions: Other: Comparator arm

INTERVENTIONS:
Other: FIT Plus — * Group handwashing facilities
  * Daily group handwashing and toothbrushing activities
  * Sanitation operation and maintenance manuals for school officials
  * Toilet cleaning consumable
  * Toilet and handwashing station maintenance kits
  * Soap, toothbrushes, and toothpaste
  Arms: Fit Plus
Other: Comparator arm — This is the same intervention as FIT Plus, but will be delivered to schools following endline data collection
  Arms: Comparator

SUMMARY:
This study will assess the impact of a school-based water, sanitation, and hygiene management intervention on toilet use and pupil handwashing in the Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Attending study school on day of observation

Exclusion Criteria:

* No predefined exclusion criteria since individual-level data is not recorded.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8687 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Toilet Usability Index | 5 months after intervention delivery
  The Toilet Usability Index is a composite score based on toilet availability, accessibility, and privacy collected through direct observation of facilities.

SECONDARY OUTCOMES:
Soap Use Ratio | 5 months after intervention delivery
  The secondary outcome measure is the soap-use ratio per toilet, which will be calculated based on the weight of soap used in one day divided by the number of toileting events in the same day.

CONTACTS AND LOCATIONS:
Locations (1):
- GIZ / Fit For School, Manila, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buxton H, Dimaisip-Nabuab J, Duijster D, Monse B, Benzian H, Dreibelbis R. The impact of an operation and management intervention on toilet usability in schools in the Philippines: a cluster randomised controlled trial. BMC Public Health. 2019 Dec 16;19(1):1680. doi: 10.1186/s12889-019-7833-7. PMID 31842809